CLINICAL TRIAL: NCT04988672
Title: OPTIMISER Registry - A Prospective Cohort Study to Describe the OPTIMal Management and Outcomes of PatIents PreSEnting With Acute MyocaRdial Infarction
Acronym: OPTIMISER
Status: Recruiting | Type: Observational
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Matthias Bossard, Co-principal Investigator, Luzerner Kantonsspital
Other Study IDs: 2020-02559
Record Dates: First submitted 2021-07-25; First posted 2021-08-03 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Myocardial Infarction; Myocardial Ischemia; STEMI; NSTEMI
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the OPTIMISER Registry is to prospectively and retrospectively collect baseline, clinical and procedural data in patients who present with AMI and are treated with PCI as well as prospectively collect the clinical outcome data. Outcomes will be compared in different clinical subgroups. The impact of PCI in AMI in general as well as cardiovascular outcomes after AMI will be assessed.

DETAILED DESCRIPTION:
* To assess procedural success and clinical outcomes among persons with AMI, who undergo PCI and/ or CABG for AMI (STEMI or NSTEMI)

  1. Periprocedural outcomes/ complications, which will be analyzed, represent: final result (e.g. TIMI flow), stent expansion, dissections, perforations, prevalence of thrombus (assessed by angiography and intravascular imaging)
  2. Short and long-term clinical outcomes of interest including: new AMI, unstable angina (UA), stent-/scaffold thrombosis, target lesion failure, target vessel revascularization, ischemia driven revascularization, repeat hospitalization, new/worsening heart failure, cardiogenic shock, stroke, bleedings, cardiovascular death and all-cause death.
* To describe procedural and clinical performance of various balloon, stent and scaffold devices implanted in patients presenting with AMI during the afore mentioned period
* To study the impact of different devices and strategies used for lesion preparation and PCI optimization strategies among patients undergoing PCI
* To describe early and late angiographic and OCT-findings among coronary artery disease in patients with AMI treated with various metallic stent and scaffold devices
* To assess possible predictors for coronary stent implantation or device failure
* To evaluate the impact of different antithrombotic regimens on patient clinical outcomes
* To study procedural and clinical outcomes among CAD patients requiring hemodynamic support using mechanical devices.
* To describe economic implications (cost-effectiveness) of various interventional treatments for CAD.

ELIGIBILITY:
Inclusion Criteria:

* Subject >18 years of age
* Individuals who are newly diagnosed with AMI or have been diagnosed with AMI (STEMI or NSTEMI) within the last 5 years (since 2016).
* Subjects must be willing to sign a patient informed consent (PIC) OR a patient ́s relative/ proxy are willing to provide PIC or patients have signed the General Consent (GK).

Exclusion Criteria:

* Patient unwilling or unable to provide informed consent
* Patients with no ACS/AMI (e.g. Takotsubo cardiomyopathy, acute heart failure not related to AMI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In an all-comers design, virtually any AMI patient treated with PCI or CABG at the Cardiology Division of Lucerne Cantonal Hospital and giving consent may be included. We expect a total inclusion rate of around 400 patients per year at the LUKS. The prospective recruitment is planned to continue for 10 years, which results in 4000 patients in the prospective arm. In addition, a retrospective arm will include a random sample of 500 patients who presented with AMI and were treated with PCI or CABG in the 5 years prior to study start (2016-2020).
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of major adverse cardiac and cerebrovascular events (MACCE) (including new AMI, stroke or cardiovascular death) at 1 year | at 1 year

SECONDARY OUTCOMES:
Rate of major adverse cardiac and cerebrovascular events (MACCE) | 1, 2, 5 and 10 years
Rate of new AMI | 1, 2, 5 and 10 years
Rate of TIA or stroke | 1, 2, 5 and 10 years
Rate of stent thrombosis | 1, 2, 5 and 10 years
Rate of target vessel revascularization | 1, 2, 5 and 10 years
Rate of target lesion failure | 1, 2, 5 and 10 years
Rate of ischemia-driven revascularization | 1, 2, 5 and 10 years
Rate of unstable angina | 1, 2, 5 and 10 years
Rate of rehospitalization for recurrent angina | 1, 2, 5 and 10 years
Rate of hospitalization for heart failure | 1, 2, 5 and 10 years
Rate of rehospitalisation for heart failure, resuscitated cardiac arrest or implantable cardioverter-defibrillator (ICD) implantation at follow- up. | 1, 2, 5 and 10 years
Rate of cardiovascular mortality | 1, 2, 5 and 10 years
Rate of all-cause mortality | 1, 2, 5 and 10 years
Rate of bleeding events (access site or non-access site related) according to the BARC classification. | 1, 2, 5 and 10 years
Rate of vascular complications (according to VARC criteria) | 1, 2, 5 and 10 years
Rate of new York Heart Association (NYHA) class | 1, 2, 5 and 10 years
Rate of cardiogenic shock | 1, 2, 5 and 10 years
Rate of acute renal failure | 1, 2, 5 and 10 years
Rate of new atrial fibrillation | 1, 2, 5 and 10 years
Rate of new ventricular arrhythmias | 1, 2, 5 and 10 years
Rate of major adverse limb events (MALE) | 1, 2, 5 and 10 years
Rate of periprocedural complications (e.g. coronary perforations, no- reflow) | 1, 2, 5 and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Florim Cuculi, M.D., Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Heart Centre, Lucerne, Switzerland

REFERENCES:
- [Background] Tersalvi G, Attinger-Toller A, Kalathil D, Winterton D, Cioffi GM, Madanchi M, Seiler T, Stadelmann M, Goffredo F, Fankhauser P, Moccetti F, Wolfrum M, Toggweiler S, Bloch A, Kobza R, Cuculi F, Bossard M. Trajectories of Cardiac Function Following Treatment With an Impella Device in Patients With Acute Anterior ST-Elevation Myocardial Infarction. CJC Open. 2022 Nov 5;5(1):77-85. doi: 10.1016/j.cjco.2022.11.002. eCollection 2023 Jan. PMID 36700188
- [Background] Cioffi GM, Madanchi M, Bossard M, Cuculi F. Deferring stent optimization in stent thrombosis: A novel approach for STEMI management-Insights from a case series. Clin Case Rep. 2021 Feb 13;9(3):1150-1154. doi: 10.1002/ccr3.3697. eCollection 2021 Mar. PMID 33768799